CLINICAL TRIAL: NCT03110146
Title: EnSite Precision 2.1 Feasibility Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10173
Record Dates: First submitted 2017-02-02; First posted 2017-04-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EnSite Precision — Ablation procedure

SUMMARY:
The objective is to demonstrate feasibility of new 'Magnetic Primary' catheter tracking algorithms within the Velocity Research Platform (VRP) by assessing the frequency of shift/drift during ablation compared to the current commercial EnSite Precision 2.0.1

The secondary objective is to evaluate catheter rendering in the VRP system.

DETAILED DESCRIPTION:
This is an acute, multi-center, observational, prospective feasibility study with up to 80 patients at up to 5 centers in Europe.

Data will be simultaneously collected on both the EnSite Precision 2.0.1 and VRP mapping systems for the entire duration of the EP mapping and ablation procedure. This study will not require significant change to the current clinical workflow of the mapping and ablation procedure. The VRP operator will observe both displays in real-time and will enter extensive electronic annotations to the VRP data stream to facilitate retrospective analysis. Examples of annotations include drug administration, patient movement, and the introduction of devices such as an intracardiac Echography (ICE) catheter which are not visible on the EnSite mapping system.

If/when the VRP operator notices events which might be better understood with additional data, he/she might ask the physician to hold a catheter in a stable position for an extra few seconds and/or move the catheter to another position. Examples of such events include catheters appearing outside the 3D model and unrealistic catheter shapes on either display. Compliance with such requests is optional and subject to physician preference.

Retrospective data analysis will focus on characterization of the following:

* Occurence rates and potential causes for Shift and Drift.
* Frequency and severity of discrepancies between impedance and magnetic coordinates.
* Positions of catheters relative to the 3D model.
* Positions of catheters relative to each other, comparing to fluoroscopic images when available.
* Shapes of catheters on the research system as the catheters are moved to different locations.
* Final geometry apprearance on the VRP.
* Voltage and timing maps appearance on the VRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for a cardiac EP study and ablation procedure using a 3D mapping system.
* Over 18 years of age
* Ability to provide informed consent for study participation and be willing and able to comply with the protocol described evaluations.

Exclusion Criteria:

* Pregnant or possibly pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing a cardiac EP mapping and ablation procedure in which a SJM sensor-enabled catheter and the EnSite Precision Cardiac Mapping system is used, is considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Demonstrate feasibility of new algorithms witihn the EnSite Velocity Research Platform (VRP) by assessing the frequency of shift/drift during ablation compared to the current commercial EnSite Precision 2.0.1. | Up to 12 months
  Demonstrate feasibility of new algorithms within the EnSite Velocity Research Platform (VRP) by assessing the frequency of shift/drift during ablation compared to the current commercial EnSite Precision 2.0.1

IPD SHARING:
Plan to Share IPD: Undecided